CLINICAL TRIAL: NCT00363714
Title: A Dose Escalation Trial of an Intravitreal Injection of Sirna-027 in Patients With Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: Sirna Therapeutics Inc. (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIRNA 0401; AGN211745; NCT00495742 (obsolete NCT alias)
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Age-Related Macular Degeneration; Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

ARMS (6):
- 1 (Experimental): Single intravitreal injection
  Interventions: Drug: AGN211745
- 2 (Experimental): Single intravitreal injection
  Interventions: Drug: AGN211745
- 3 (Experimental): Single intravitreal injection
  Interventions: Drug: AGN211745
- 4 (Experimental): Single intravitreal injection
  Interventions: Drug: AGN211745
- 5 (Experimental): Single intravitreal injection
  Interventions: Drug: AGN211745
- 6 (Experimental): Single intravitreal injection
  Interventions: Drug: AGN211745

INTERVENTIONS:
Drug: AGN211745 — 100microgram single intravitreal injection
  Other Names: Sirna-027
  Arms: 1
Drug: AGN211745 — 200microgram single intravitreal injection
  Other Names: Sirna-027
  Arms: 2
Drug: AGN211745 — 400microgram single intravitreal injection
  Other Names: Sirna-027
  Arms: 3
Drug: AGN211745 — 800microgram single intravitreal injection
  Other Names: Sirna-027
  Arms: 4
Drug: AGN211745 — 1200microgram single intravitreal injection
  Other Names: Sirna-027
  Arms: 5
Drug: AGN211745 — 1600microgram single intravitreal injection
  Other Names: Sirna-027
  Arms: 6

SUMMARY:
The purpose of this study will be to assess the safety and tolerability and dose-limiting toxicity of a single intravitreal injection of Sirna-027 (AGN211745) and to assess the anatomical changes in the retina, changes in CNV, and changes in visual acuity. Escalation to the next dose cohort will be completed following minimum of 2 weeks follow-up. Patients will be monitored intensively for three months, and then followed-up for safety up to 24 months post-injection.

ELIGIBILITY:
Inclusion Criteria:

* Active AMD with Subfoveal CNV (classic and/or occult CNV)
* CNV lesion thickness >/= 250um by OCT assessment
* Visual acuity in study eye of </= 20/100 but not worse than 20/800
* Not eligible for or refused standard treatment

Exclusion Criteria:

* Females of childbearing potential
* Other causes of CNV including pathologic myopia, the ocular histoplasmosis syndrome, angioid streaks, choroidal rupture and multifocal choroiditis
* Any intraocular surgery or treatment of AMD with Visudyne within 3 months of study entry
* CNV lesion >/= 12 MPS disc area

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Time frame 3 months: Baseline/Day 1, Day 2, Day 7, Day 14, Day 28, Day 56, Day 84

SECONDARY OUTCOMES:
Visual Acuity using the Diabetic Retinopathy Study chart | Time frame 24 months: Screening, Day 1, Day 2, Day 7, Day 14, Day 28, Day 56, Day 84, Month 6, Month 9, Month 12, Month 18, Month 24
IOP | Time frame 24 months: Screening, Day 1, Day 2, Day 7, Day 14, Day 28, Day 56, Day 84, Month 6, Month 9, Month 12, Month 18, Month 24
OCT | Time frame 3 months: Screening, Day 7, Day 14, Day 28, Day 56, Day 84
Fluorescein Angiography (FA) | Time frame 24 months (Screening, Day 7, Day 14, Day 28, Day 84 and Month 24)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- United States (2):
  - Baltimore, Maryland
  - Cleveland, Ohio

REFERENCES:
- [Derived] Kaiser PK, Symons RC, Shah SM, Quinlan EJ, Tabandeh H, Do DV, Reisen G, Lockridge JA, Short B, Guerciolini R, Nguyen QD; Sirna-027 Study Investigators. RNAi-based treatment for neovascular age-related macular degeneration by Sirna-027. Am J Ophthalmol. 2010 Jul;150(1):33-39.e2. doi: 10.1016/j.ajo.2010.02.006. PMID 20609706